CLINICAL TRIAL: NCT06315062
Title: Efficacy of Rezum® in Reducing Prostate Volume. A Retrospective Study in Patients With Benign Hyperplasia in Costa Rica
Brief Title: Efficacy of Rezum® in Reducing Prostate Volume
Status: Completed | Type: Observational
Sponsor: Urología Costa Rica (Other)
Responsible Party: Principal Investigator, Mario González, Principal Investigator, Urología Costa Rica
Other Study IDs: CEC-UNIBE-07-2023
Record Dates: First submitted 2024-02-22; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Benign Hyperplasia of Prostate
Keywords: Prostate; Urology; IPSS score; clinical efficacy; Rezum
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to assess the efficacy of Rezum® water vapor therapy in reducing prostate volume in patients aged 40 years or older with Benign Prostate Hyperplasia (BPH) at UNIBE Hospital in Costa Rica. A retrospective analysis will be conducted on 289 patient records, focusing on prostate volume, International Prostate Symptom Score (IPSS), and urinary flow rate. Statistical analyses included two-sample mean comparisons, effect size estimation, and linear regression.

DETAILED DESCRIPTION:
Abstract:

Aim

To estimate the effect size of the prostate volume reduction after application of water vapor injections (Rezum®) in 40 years or older patients, that have been diagnosed with Benign Prostate Hyperplasia (BPH) and are registered at UNIBE Hospital. This contrast provides a retrospective efficacy of the minimally invasive treatment valid for the local population.

Methods:

A retrospective study will be conducted to review patient records, attended at UNIBE Hospital, in Costa Rica. Prostate volume was established as the main variable to assess BPH reversion. Other variables like the International Prostate Symptome Score (IPSS) and urinary flow rate were also evaluated for each patient.

Two sample mean comparisons of baseline and follow up measures for prostate volume and IPSS will be calculated to estimate a mean difference. Effect size parameters like Cohen's d, Hedges's g and Glass's delta were also estimated and compared based on the standard deviation assessment. A linear regression model will also adjuste to obtain values of the statistical contribution from each of the variables included to evaluate the clinical reversal of a benign prostate hyperplasia diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Men who received Rezum therapy
* Men who have been treated at the UNIBE Hospital in Urology by Dr. González

Exclusion Criteria:

* Patients without complete data for the previous variables

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records of people who have been urology consultants and treated by Dr. Mario González Salas at the UNIBE Hospital from 2020 to the present.
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Prostate volume | at 0, 1, 3 and 6 months.
  Prostate volume

SECONDARY OUTCOMES:
International Prostate Symptome Score | at 0, 1, 3 and 6 months.
  International Prostate Symptome Score, minimun score is 0 with midly simptomatic and 35 is the maximun value meaning severely symptomatic
Urinary flow rate | at 0, 1, 3 and 6 months.
  Urinary flow rate

CONTACTS AND LOCATIONS:
Overall Officials: Mario González Salas, Dr., Principal Investigator — Hospital UNIBE; Milena Castro Mora, PhD., Study Director — Universidad de Costa Rica
Locations (1):
- Hospital UNIBE, San José, Costa Rica